CLINICAL TRIAL: NCT02505737
Title: Improving Access to Depression Care in Parkinson's Disease: A Telehealth Approach
Brief Title: Telephone-Based Counseling for Depression in Parkinson's Disease
Acronym: TH-CBT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: Michael J. Fox Foundation for Parkinson's Research (Other)
Responsible Party: Principal Investigator, Roseanne D Dobkin, PhD, Associate Professor of Psychiatry, Rutgers, The State University of New Jersey
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20150001714
Record Dates: First submitted 2015-07-21; First posted 2015-07-22 (Estimated); Last update posted 2019-02-19 (Actual); Status verified 2019-02

CONDITIONS: Depression; Parkinson's Disease
MeSH Terms: conditions — Depression; Parkinson Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- TH-CBT (Experimental): The treatment works by teaching people with PD (PWP) the coping skills needed to manage their emotional reactions to the numerous challenges posed by the disease. Specifically, the treatment targets maladaptive thought patterns (e.g., I have no control; I am helpless) and behaviors (e.g., social isolation, lack of exercise, poor sleep habits, excessive worry), and critically, provides caregivers with the tools needed to encourage the PWPs' practice of their newly acquired coping skills. Treatment is administered over the phone and no travel is required.
  Interventions: Behavioral: TH-CBT
- Enhanced Usual Care (Other): All participants will continue to receive their routine medical treatment under the supervision of their personal doctors (e.g., neurologists, psychiatrists, primary care physicians, therapists) while participating in the study. This routine treatment (e.g., usual care) will be further enhanced with the provision of written educational materials for effective coping with PD, the close clinical monitoring of depressive symptoms by study staff, and the provision of counseling resources in the local community.
  Interventions: Other: Enhanced Usual Care

INTERVENTIONS:
Behavioral: TH-CBT — Telephone-Based Cognitive Behavioral Therapy (TH-CBT). A 10-session treatment protocol that incorporates behavioral activation, thought monitoring and restructuring, relaxation training, worry control, sleep hygiene, and caregiver psychoeducation and support
  Arms: TH-CBT
Other: Enhanced Usual Care — Community-based treatment as usual and supplemental reading material
  Arms: Enhanced Usual Care

SUMMARY:
There is a critical need for treatments that address depression and barriers to mental health care in Parkinson's disease (PD). This randomized-controlled trial will evaluate a 10-session telephone-guided cognitive behavioral self-help program (TH-CBT) for depression in PD (dPD). 72 people with dPD (and their caregivers) will receive either TH-CBT plus enhanced usual care (INTERVENTION GROUP) or enhanced usual care only (CONTROL GROUP). Groups will be compared at baseline, midpoint, endpoint, and 1 and 6 months post-treatment. Participants assigned to the control group with have the opportunity to receive the experimental intervention (TH-CBT) after the data collection period (e.g., after the 6-month follow-up evaluation). Given the public health impact of improved depression treatment in PD, the knowledge to be gained may be significant and the project could directly impact clinical practice.

DETAILED DESCRIPTION:
All study procedures, including the initial evaluation, study treatment sessions, and follow-up study assessments, take place over the phone and no travel is required. All PWP across the USA may participate.

All participants will continue to receive their routine medical treatment under the supervision of their personal doctors (e.g., neurologists, psychiatrists, primary care physicians, therapists) while participating in the study. In addition to usual care, half of the participants in the study will receive the experimental telehealth treatment (TH-CBT; intervention group), immediately after enrolling in the research program. The other half will only receive usual care (control group) and will have the option to receive TH-CBT, after completing all study related assessments (9 months after the initial evaluation). Group assignment will be decided randomly (i.e., by chance).

Study eligibility will be determined by a qualified professional. Those who qualify for participation will be randomly assigned (e.g., flip of a coin) to either the intervention (TH-CBT) or the control group (enhanced usual care).

Participants assigned to the TH-CBT group will receive a 10-chapter CBT self-help treatment workbook, tailored to the unique needs of people with PD, immediately following enrollment. Participants will read and complete one treatment module per week (approximately 60 minutes per module plus practice exercises throughout the week). The treatment materials will review different coping skills for the effective management of depression. Study therapists will call participants to review the treatment material over the phone every week (after every chapter) or every other week (after ever 2 chapters), based on participant needs. These telephone-based counseling sessions will last 60 minutes. It will take approximately 10 weeks to complete the study treatment materials.

A family member or friend (carepartner) will also be asked to participate in 3-4 separate educational sessions (30-60 minutes each), evenly dispersed throughout the 10 week TH-CBT treatment period. The study treatment provided to the care-partner will teach the care-partner how to best support the participant with PD as he/she tries to incorporate the information learned during the study treatment, in day-to-day life.

Participants will be re-evaluated 6, 11, 15, and 35 weeks after the initial evaluation.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed diagnosis of Parkinson's disease.
2. Clinically significant depressive symptoms (e.g., symptoms are pervasive, distressing, and make life harder). The presence of a formal depressive disorder will be determined by study staff based on standardized criteria (e.g., SCID).
3. 35-85 years old
4. Stable medication regimen ≥ 6 weeks
5. No change in mental health treatment in the past 2 months
6. Family member or friend willing to participate
7. Access to a telephone
8. Live in the United States of America (USA)

Exclusion Criteria:

1. Suicidal plans or intent
2. Probable Dementia or Significant Cognitive Impairment
3. Significant motor fluctuations (i.e., ≥ 50% of the day)
4. Unstable medical conditions
5. Bipolar, Psychotic Spectrum, or Substance Abuse Disorders

Ages: 35 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
Depression on the Hamilton Depression Rating Scale | 9 months
  clinician-administered scale- depression

SECONDARY OUTCOMES:
Treatment Response on the Clinical Global Impression- Improvement Scale | 9- months
  clinician-administered scale- treatment response
Anxiety on the Hamilton Anxiety Rating Scale | 9-months
  clinician administered scale-anxiety
Quality of life on the SF-36 | 9-months
  self-report scale- quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Roseanne D Dobkin, PhD, Principal Investigator — Rutgers Robert Wood Johnson Medical School
Locations (1):
- Rutgers University-Robert Wood Johnson Medical School, Piscataway, New Jersey, United States

REFERENCES:
- [Derived] Dobkin RD, Mann SL, Gara MA, Interian A, Rodriguez KM, Menza M. Telephone-based cognitive behavioral therapy for depression in Parkinson disease: A randomized controlled trial. Neurology. 2020 Apr 21;94(16):e1764-e1773. doi: 10.1212/WNL.0000000000009292. Epub 2020 Apr 1. PMID 32238507